CLINICAL TRIAL: NCT05798195
Title: Traditional Chinese Medicine or Low-dose Dexamethasone in Symptomatic Patients With Post-COVID-19 Parenchymal Lung Abnormalities: a Randomized Controlled Trial Three Arm, Parallel Group, Single Blind, Randomized Controlled Trial.
Brief Title: Traditional Chinese Medicine or Low-dose Dexamethasone in COVID-19 Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Chief physician of PCCM, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-ZF-3
Record Dates: First submitted 2023-04-02; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- controlled group (Active Comparator): conventional western medicine treatment including oxygen therapy, antibiotics, nebulization therapy, etc.
  Interventions: Other: conventional western medicine treatment
- dexamethasone group (Experimental): dexamethasone 1.5mg/day for one week and 0.75mg/day for another week basing on conventional western medicine.
  Interventions: Other: conventional western medicine treatment; Drug: Dexamethasone oral tablet
- Chinese medicine group (Experimental): Strengthening spleen and tonifying lung decoction for 2 weeks basing on conventional western medicine.
  Interventions: Other: conventional western medicine treatment; Other: Traditional Chinese medicine decoction

INTERVENTIONS:
Other: conventional western medicine treatment — conventional western medicine treatment only
Drug: Dexamethasone oral tablet — treat with Dexamethasone for 2 weeks
  Arms: dexamethasone group
Other: Traditional Chinese medicine decoction — treat with strengthening spleen and tonifying lung decoction for 2 weeks
  Arms: Chinese medicine group

SUMMARY:
The goal of this type of clinical trial is to learn about symptomatic patients with post-COVID-19 parenchymal lung abnormalities. The main questions it aims to answer are: the efficacy and safety of low-dose dexamethasone or traditional Chinese medicine in symptomatic patients with post-COVID-19 parenchymal lung abnormalities.

Participants will be divided into three parallel groups：controlled group with conventional western medicine treatment including oxygen therapy, antibiotics, nebulization therapy, etc. dexamethasone group: dexamethasone 1.5mg/day for one week and 0.75mg/day for another week basing on conventional western medicine. Chinese medicine group: Strengthening spleen and tonifying lung decoction for 2 weeks basing on conventional western medicine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COVID-19 pneumonia；
* 3 to 8 weeks after the onset of the first symptoms of COVID-19 infection;
* Modified Medical Research Council (mMRC) score ⩾2 or hypoxemia;
* Imaging severity assessment of pneumonia: CT severity scores (CTSS):≥5；
* Signed the informed consent.

Exclusion Criteria:

* Participants still admitted to intensive care unit at the time of enrollment;
* Known prior structural lung disease, including pulmonary fibrosis, severe COPD, severe bronchiectasis, and lung destruction;
* Taking glucocorticoids or immunosuppressants because of other chronic diseases;
* Contraindications of glucocorticoid;
* Heart failure(NYHA III or IV);
* Participants with renal replacement therapy;
* Psychiatric disorders or cognitive impairments;
* The expected survival time is less than six months due to diseases other than COVID-19 pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung CT scan | 1 month
  compared with base,≥90% pneumonia obsorbed

SECONDARY OUTCOMES:
Lung CT scan | 3 months
  compared with base,≥50% pneumonia obsorbed

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Zhai, Dcotor, Principal Investigator — Department of Respiratory and Critical Care Medicine
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China